CLINICAL TRIAL: NCT00919737
Title: A Phase 1/2, Multicenter, Non-Randomized, Open Label Clinical Trial of NPC-08 Implant in Patients Undergoing Surgery for Newly-Diagnosed Malignant Glioma and Recurrent Glioblastoma Multiforme.
Brief Title: Study of NPC-08 is to Treat for Newly-Diagnosed Malignant Glioma and Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-08-1
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Malignant Glioma
Keywords: NPC-08; carmustine; nitrosourea; safety
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NPC-08 (Experimental)
  Interventions: Drug: NPC-08

INTERVENTIONS:
Drug: NPC-08 — Polifeprosan 20 with Carmustine 3.85%

SUMMARY:
The purpose of this study is to evaluate whether NPC-08 is safety and efficacy in the treatment of newly-diagnosed malignant glioma and recurrent glioblastoma multiforme.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged between 18 and 65 years;
* Radiographic evidence on cranial MRI of a single contrast-enhancing unilateral supratentorial cerebral tumor;
* Karnofsky Performance Score of 60 or higher;
* Willing to practice an effective method of birth control for at least 12 months after wafer implantation surgery;

Exclusion Criteria:

* More than one focus of tumor or tumor crossing the midline, as assessed by coronal cranial MRI scan;
* Prior radiotherapy to the brain;
* Prior chemotherapy for the malignant glioma before the baseline evaluation, or patients who were being treated with chemotherapeutic agents;
* Known hypersensitivity to nitrosoureas;
* Participation in any other investigational protocol in the previous 6 months for any type of malignancy;

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Overall survival to 12 months | 12 months

SECONDARY OUTCOMES:
Progression-free survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Masao Mastutani, M.D., D.M.Sci., Study Director — Saitama International Medical Center, Saitama Medical University
Locations (1):
- The Tazuke Kofukai Foundation Medical Research Kitano Hospital, Osaka, Osaka, Japan